CLINICAL TRIAL: NCT01656330
Title: Randomized, Parallel-Group, Open-Label Study to Assess the Effects of 3-Factor and 4-Factor Prothrombin Complex Concentrates on the Pharmacodynamics of Rivaroxaban
Brief Title: A Study to Assess the Effects of 2 Different Prothrombin Complex Concentrates on the Pharmacodynamics of Rivaroxaban in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR100867; RIVAROXNAP1003 (Other: Janssen Pharmaceutical Research & Development, LLC); 2012-002313-20 (EudraCT Number)
Record Dates: First submitted 2012-07-31; First posted 2012-08-03 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Healthy; Rivaroxaban; JNJ-39039039; BAY59-7939; Prothrombin Complex Concentrate (PCC)
MeSH Terms: conditions — Hemophilia B | interventions — Rivaroxaban; Profilnine SD; factor IX, factor VII, factor X, prothrombin drug combination; Sodium Chloride

ARMS (3):
- Rivaroxaban + Profilnine SD (Experimental): Rivaroxaban 20 mg twice a day on Days 1-4 followed by rivaroxaban 20 mg once a day on Day 5 administered 4 hours before a single bolus dose of Profilnine SD 50 IU/kg.
  Interventions: Drug: Rivaroxaban 20 mg twice daily; Drug: Rivaroxaban 20 mg once daily; Drug: Profilnine SD
- Rivaroxaban + Beriplex P/N (Experimental): Rivaroxaban 20 mg twice a day on Days 1-4 followed by rivaroxaban 20 mg once a day on Day 5 administered 4 hours before a single bolus dose of Beriplex 50 IU/kg.
  Interventions: Drug: Rivaroxaban 20 mg twice daily; Drug: Rivaroxaban 20 mg once daily; Drug: Beriplex P/N
- Rivaroxaban + Saline (Experimental): Rivaroxaban 20 mg twice a day on Days 1-4 followed by rivaroxaban 20 mg once a day on Day 5 administered 4 hours before a single 100cc bolus of saline.
  Interventions: Drug: Rivaroxaban 20 mg twice daily; Drug: Rivaroxaban 20 mg once daily; Other: Saline

INTERVENTIONS:
Drug: Rivaroxaban 20 mg twice daily — One rivaroxaban 20 mg tablet administered twice a day (b.i.d.) for 4 days (Days 1-4). Interpretation by CTRL: Concentration type = Exact; Number = 20; unit=mg; route: oral use for 4 days.
Drug: Rivaroxaban 20 mg once daily — One rivaroxaban 20 mg tablet administered once daily on Day 5. Interpretation by CTRL: Concentration type = Exact; Number = 20; unit=mg; route: oral use for 1 day.
Drug: Profilnine SD — Single bolus dose of Profilnine SD 50 IU/kg administered by intravenous (IV) injection on Day 5. Interpretation by CTRL: Concentration type = Exact; Number = 50; unit=IU/kg; route: intraveous use.
  Arms: Rivaroxaban + Profilnine SD
Drug: Beriplex P/N — Single bolus dose of Beriplex P/N 50 IU/kg administered by intravenous (IV) injection on Day 5 Interpretation by CTRL: Concentration type = Exact ; Number = 50; unit=IU/kg; route : intravenous use
  Arms: Rivaroxaban + Beriplex P/N
Other: Saline — Single 100 cc bolus of saline administered by intravenous (IV) injection on Day 5. Interpretation by CTRL: Concentration type = Exact ; Number = 100; unit=cc; route : intravenous use use.
  Arms: Rivaroxaban + Saline

SUMMARY:
The purpose of this study is to assess the use of 2 different Prothrombin Complex Concentrates (PCCs) on their ability to reverse (normalize) the pharmacodynamic effects of rivaroxaban in healthy adult volunteers.

DETAILED DESCRIPTION:
This is a single-center, open-label (volunteers and staff will know the identity of all treatments), randomized (volunteers assigned to treatment by chance) study in healthy adult volunteers to assess the effects of 2 different Prothrombin Complex Concentrates (PCCs) (drugs that act to control bleeding) on the pharmacodynamics (ie, the study of the biochemical and physiological effects of a drug on the body) of rivaroxaban (a drug that acts to prevent the formation of blood clots). Eligible volunteers will receive treatment with rivaroxaban administered orally (by mouth) on Days 1-4. On Day 5, rivaroxaban will be administered orally before the randomized intravenous (IV) (into the vein) administration of 1 of 3 treatments: Profilnine SD (a 3-factor PCC), Beriplex P/N (a 4-factor PCC), or saline. Blood samples will be collected from healthy volunteers during the study to assess the activity of rivaroxaban. Safety will be monitored throughout the study. The total length of participation in the study for each volunteer will be approximately 28 days (includes a 21-day Screening Period and a 7-day Treatment Period).

ELIGIBILITY:
Inclusion Criteria:

* Have coagulation test results of PT, INR and aPTT that are within normal limits
* Have a Body Mass Index (BMI; weight [kg]/height2 [m]2) between 18 and 30 kg/m2 (inclusive), and body weight between 50 and 100 kg
* Have blood pressure (after the volunteer is supine [lying down with the face up] for 5 minutes) between 90 and 140 mmHg systolic, inclusive, and between 50 and 90 mmHg diastolic
* Non-smoker

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic (blood) disease, thrombosis, coagulation (blood clotting) disorders, lipid abnormalities, significant pulmonary (lung) disease, diabetes mellitus, renal (kidney) or hepatic (liver) insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the volunteer or that could interfere with the interpretation of the study results
* History of serious bleeding in the past, including gastrointestinal bleeding requiring hospitalization, intracranial (in the brain) bleeding of any type, or uncontrollable postoperative bleeding
* History of intracranial tumor or aneurysm or known abdominal aneurysm
* Known allergy to the study drug or any of the excipients of the formulation
* Known allergy to heparin or history of heparin-induced thrombocytopenia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Measurement of pharmacodynamic (PD) variables: prothrombin time (PT), International Normalized Ratio (INR), activated partial thromboplastin time (aPTT), thrombin generation assay (TGA) and anti-Factor Xa (anti-FXa) | Days 1-6
  Pharamacodymic (PD) variables (ie, PT, INR, aPTT, TGA, and anti-FXa) are blood coagulation (or clotting) tests. These blood clotting tests will be performed to assess the effects of Prothrombin Complex Concentrates (PCCs) (Profilnine SD or Beriplex P/N) on the pharmacodynamics of rivaroxaban.

SECONDARY OUTCOMES:
Rivaroxaban plasma concentrations | Days 1-6
  Rivaroxaban plasma concentrations will be measured to assess the pharmacokinetics (the study of the extent and rate of absorption, distribution, metabolism, and excretion of a drug in the body [ie, the study of what the body does to the drug]) of rivaroxaban at steady state (steady state is the time when the rate of absorption of the drug into the body equals the rate of elimination from the body).
The number of healthy volunteers reporting adverse events | Days 1-6
  Adverse events reported are used to assess the safety and tolerability of study drugs.
Changes from baseline in clinical laboratory tests performed | Day 1; Day 6
  Clinical laboratory tests include chemistry, hematology, urinalysis, and coagulation. Baseline for all laboratory evaluations will be defined as the last evaluation done before the first study drug administration.
Change from baseline in electrocardiogram (ECG) findings | Day 1; Day 6
  Baseline for all ECG measurements will be defined as the last evaluation done before the first study drug administration.
Change from baseline physical examination findings | Day 1; Day 6
  Baseline for all physical examinations will be defined as the last evaluation done before the first study drug administration.
Change from baseline in vital signs measurements | Day 1; Day 6
  Vital signs measurements include pulse/heart rate and blood pressure (systolic and diastolic). Baseline vital signs measurements will be defined as the last evaluation done before the first study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, L.L.C Clinical Trial, Study Director — Janssen Research & Development, L.L.C
Locations (1):
- Merksem, Belgium